CLINICAL TRIAL: NCT04703907
Title: Auricular Stimulation (AS) vs. "Waiting List" for Relief of Stress and Anxiety in Health Care Workers During COVID-19 Pandemic - a Prospective Controlled Investigation
Brief Title: Auricular Stimulation for Relief of Stress and Anxiety
Acronym: AA_COVID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BB 324/20
Record Dates: First submitted 2021-01-08; First posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Stress and Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Prospective investigation during 15 weeks of treatment for each participant with "waiting list" control group (no intervention). Waiting group will receive the intervention (auricular stimulation) after 15 weeks of investigation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This group is constituted from patients who will receive the intervention first within 15 weeks
  Interventions: Other: Auricular stimulation
- Waiting list (No Intervention): This group is constituted from patients who will receive the intervention after 15 weeks

INTERVENTIONS:
Other: Auricular stimulation — Auricular "acupuncture-like" stimulation (percutaneous sensory stimulation of cranial nerves)
  Arms: Intervention group

SUMMARY:
The aim of the study is to evaluate whether auricular stimulation (percutaneous sensory stimulation of cranial nerves) as compared vs. no intervention (waiting list) reduces stress and anxiety in health care providers, working at the time of COVID-19 pandemic at the University Medicine of Greifswald.

ELIGIBILITY:
Inclusion Criteria:

1. Medical care workers at the University Medicine of Greifswald
2. Experiencing stress and anxiety in connection with COVID-19 pandemic
3. Participants without previous anxiolytic medication
4. Ability to understand and fill in the structured questionnaire (Appendix D & E)
5. Written informed consent

Exclusion Criteria:

1. Recidivist alcoholics
2. Local auricular skin infection
3. Pregnant or lactating women
4. Participants with prosthetic or damaged cardiac valves and mitral valve prolaps (risk of bacterial endocarditis according to guidelines of AHA)
5. Participants who are unable to understand the consent form
6. History of psychiatric disease

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
Anxiety | 15 weeks of investigation
  State anxiety

SECONDARY OUTCOMES:
Trait anxiety | Before and after 15 weeks of intervention application
Sleep quality | 15 weeks of investigation

CONTACTS AND LOCATIONS:
Locations (1):
- University Medicine of Greifswald, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: No